CLINICAL TRIAL: NCT05798273
Title: [68Ga] Ga-PSMA-11 PET/MR-imaging of Malignant Intra-axial Brain Tumors; Primary Assessment of PSMA Expression, Optimization of Compound Delivery and Determination of Theranostic Potential
Brief Title: (68^Ga)-GaPSMA-11 PET/MR-imaging of Malignant Intra-axial Brain Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Dr. S.E.M. Veldhuijzen van Zanten, Scientific investigator, Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ErasmusMC-2020-0338
Record Dates: First submitted 2023-01-16; First posted 2023-04-04 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Malignant Brain Tumors
Keywords: Intra-axial brain tumor Malignant
MeSH Terms: interventions — Injections, Intra-Arterial

STUDY DESIGN:
Intervention Model Description: non-randomized, single center, prospective imaging study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intra-arterial injection of [68Ga]Ga-PSMA-11 (Other): eligible for intra-arterial injection (age >18 years) with enhancing glioma or brain metastases eligible for (re-)resection.
  Interventions: Procedure: intra-arterial injection; Device: synchronous PET/MRI scan; Other: Radiopharmacon Contrast agent

INTERVENTIONS:
Procedure: intra-arterial injection — All patients will receive an intravenous injection of [68Ga]Ga-PSMA-11 (1.5 MBq/kg), followed by a synchronous PET/MRI scan (median duration approximately 50 min) at 45-60 min post-injection.
  In case of a positive [68Ga]Ga-PSMA-PET signal at the tumor site, patients will return (in 2 weeks) for an intra-arterial injection (i.e., a neuro-interventional procedure) of 68Ga-PSMA-11 (1.5 MBq/kg), followed by a repeat synchronous PET/MRI scan (median duration 50 min) at 45-60 min post-injection.
Device: synchronous PET/MRI scan — Scan done at (median duration approximately 50 min) at 45-60 min post-injection.
Other: Radiopharmacon Contrast agent — Type: [68Ga]Ga-PSMA-11 dosage: 1.5 MBq/kg

SUMMARY:
PSMA is a transmembrane protein specifically expressed in the vascular endothelium of malignant brain tumors, most notably glioblastoma and not in healthy brain parenchyma. It has been shown to be involved in (neo)angiogenesis and endothelial cell invasion. By means of 68Ga-labeled PSMA ligands, investigators are able to non-invasively visualize/quantify PSMA expression in glioblastoma (neo)vasculature in vivo by means of PET.

The primary aim of this study is to confirm PSMA as suitable diagnostic and potential theranostic target in patients with intra-axial brain tumors by means of [68Ga]Ga-PSMA-HBEC-CC ([68Ga]Ga-PSMA-11) PET.

The secondary aim is to assess whether uptake is increased with intra-arterial injection in those tumors that show uptake after intravenous injection of [68Ga]Ga-PSMA-11.

DETAILED DESCRIPTION:
Brain tumors have a major impact due to both high morbidity and mortality. Primary brain tumors (glioma) have a low incidence (5-7:100,000), but the highest loss of life years compared to other cancer types. Glioblastoma without mutations in the Isocitrate Dehydrogenase gene (IDHwt), are the most frequent and the most aggressive of all primary malignant brain tumors. They account for 48% of all the primary malignant brain tumors and 15% of all primary brain tumors. Treatment consists of resection, radiotherapy and systemic chemotherapy. Nevertheless the current prognosis is still poor with a 1-, 2- and 5-year survival of respectively 40%, 17% and 6%.

Secondary brain tumors (brain metastases) are frequent, occurring in 15% of cancer patients (incidence 50-70:100,000). The prevalence of brain metastases is rising due to better extracranial local cancer control with systemic treatment resulting in more surviving patients with good local tumor control, but with brain metastases.

A recently discovered potential target for (localized) therapy of glioblastoma is PSMA. PSMA was originally found to be specifically expressed in normal prostate, and overexpressed in almost all stages of prostate cancer. In recent years, PSMA was also found to be expressed in tumor-associated (neo)vasculature in many other solid tumors, including glioblastoma.

PSMA is distinct from other vascular targets, such as vascular endothelial growth factor, endoglin, or the integrins involved in the general process of angiogenesis, as these latter are not specific to tumor vasculature. PSMA, in contrast, is not expressed in normal vasculature and is only minimally expressed in a subset of normal glial cells. PSMA therewith represents the most specific (neo)vascular target for glioblastoma currently known.

This specificity makes PSMA an ideal target for delivery of a cytotoxic agent or a radionuclide designed to tumor vasculature destruction. Particularly in intra-axial brain tumors such as glioblastoma, therapeutic targeting of (neo)vasculature is attractive as it may be exposed to a therapeutic agent much more readily than the tumor parenchyma itself, which is protected by the blood-brain barrier.

The primary aim of this first PSMA-PET study performed in the Netherlands is to confirm PSMA as suitable diagnostic and theranostic target in patients with intra-axial brain tumors by means of [68Ga]Ga-PSMA-HBEC-CC ([68Ga]Ga-PSMA-11) PET. The secondary aim is to assess whether uptake is increased with intra-arterial injection in those tumors that show uptake after intravenous injection of [68Ga]Ga-PSMA-11.

Eligible for this non-treatment study are patient, aged >18 years old, with enhancing glioma or brain metastases scheduled for (re-)resection. Upon informed consent, patients will undergo intravenous injection of [68Ga]Ga-PSMA-11, followed by synchronously combined PET-MR scans at 45-60 min post-injection to determine [68Ga]Ga-PSMA tumor uptake and dosimetry over time.

Based on the known expression profile of PSMA in glioblastoma, it is expected that significant tumor-uptake will be seen in 50% of included patients. In case the tumor shows significant uptake, patients will subsequently undergo local intra-arterial injection of [ 68Ga]GaPSMA-11, with an interval of two weeks, performed by a trained neuro-interventional radiologist, immediately followed by a repeat PET/MRI scan. Tumor uptake values of each of the scans will be compared to determine the optimal route of administration. [68Ga]Ga-PSMA-11 uptake values of the tumor will be compared to the degree of PSMA expression determined by IHC.

Based on the few studies published thus far, we expect significant expression of PSMA to be present in progressive/recurrent enhancing glioma and brain metastases. We expect approximate 50% positive scans and in these, increased uptake upon intra-arterial injection compared to intravenous injection.

The results of this pilot study will aid in the development of future PSMA-targeting chemo-

/radionuclide therapies for malignant brain tumors. Therapeutic PSMA PET imaging studies have not yet been performed in patients with primary brain tumors, but studies in patients with (cerebral) metastases from prostate cancer show promising clinical results and acceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Radiologically presumed/histologically confirmed.
* glioma (grade II-IV) showing enhancement on post-contrast MRI
* brain metastases
* Planned for (re-)resection
* Age > 18 years old
* Good clinical condition (Karnofsky performance status score >70)
* Ability and willingness to provide written informed consent

Exclusion Criteria:

* Impaired renal function: eGFR (MDRD) <30 ml/min/1,73 m2
* Impaired liver function :AST and ALT > 2.5 8 ULN
* Karnofsky Performance score of less than 70
* Previous other malignancies, except for any previous malignancy which was treated with curative intent more than 3 years prior to enrollment, and except for adequately controlled limited basal cell carcinoma of the skin, squamous carcinoma of the skin or carcinoma in situ of the cervix
* Known history of cerebrovascular disease (e.g. ischemic stroke, cerebral hemorrhage)
* Severe claustrophobia prohibiting PET/MRI scanning
* A neurologic or psychiatric condition impairing judgement, making adequate informed consent impossible
* Any psychological, familial, sociological or geographical condition hampering participation

Contra-indications for PET imaging

* Pregnancy or lactation
* Known allergic reaction to therapeutic radiopharmaceuticals
* Contra-indications for MR imaging:
* Metal implants or fragments of the type which may concentrate radiofrequency fields or cause tissue damage from twisting in a magnetic field:

  * metal plates, wires, screws or rods
  * surgical (brain) clips or staples
  * metallic fragments in or near eyes or blood vessels
  * metallic cardiac valve(s)
  * a cardiac implantable electronic device (pacemaker, wires, implantable cardioverter-defibrillator (ICD))
  * eye implants
  * ear or cochlear implants
  * a drug pump implant
  * a nerve stimulator
  * dental fillings and bridges
  * artificial joints
  * penile implants
  * tubal ligation clips
  * non-removable piercing
  * tattoos containing metal traces
* Known allergic reaction to gadolinium-based contrast agents

Contra-indications for arterial catheterization:

* Known local infection thrombus or distorted anatomy at the puncture site
* Known severe peripheral vascular disease or femoral artery disease, which makes the femoral approach impossible
* Known severe coagulopathy (spontaneous prolonged PT with an INR > 2.5)
* In case of the use of anticoagulation: an absolute contra-indication to temporarily stop or bridge the anti-coagulation.
* Known severe thrombocytopenia (platelet count 50 x 109/L)
* Allergic reaction to iodine containing contrast agent
* A physical, neurologic or psychological condition preventing the patient to lay still for the duration of the procedure (± 2h)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
tumor SUV (upon intravenous and intra-arterial injection), | 1 day
  tumor SUV (upon intravenous and intra-arterial injection
SUV tumor-to-background ratio | 1 week
  SUV tumor-to-background ratio
Biodistribution | 1 week
  Biodistribution
correlation between SUV and the degree of immunohistochemical PSMA staining | 1 week
  correlation between SUV and the degree of immunohistochemical PSMA staining

CONTACTS AND LOCATIONS:
Overall Officials: Sophie EM Veldhuijzen van Zante, Dr, Principal Investigator — Erasmus Medical Center
Locations (1):
- Laurens Groenendijk, Berkel en Rodenrijs, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pruis IJ, van Dis V, Maas SLN, Balvers RK, van den Bosch TPP, Segbers M, Veldhuijzen van Zanten SEM. PSMA radioligand uptake correlates with PSMA expression in high-grade glioma and brain metastasis: insights from a prospective PET-MRI guided multiregional biopsy study. Eur J Nucl Med Mol Imaging. 2025 Nov;52(13):4870-4881. doi: 10.1007/s00259-025-07338-4. Epub 2025 May 26. PMID 40414994